CLINICAL TRIAL: NCT03477071
Title: A 15-year Single Center Experience of Endovascular Treatment of Transplant Renal Artery Stenosis: Evaluation of Post-operative Outcomes
Brief Title: A 15-year Single Center Experience of Endovascular Treatment of Transplant Renal Artery Stenosis
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: URO-BASE03
Record Dates: First submitted 2018-03-20; First posted 2018-03-26 (Actual); Last update posted 2018-03-26 (Actual); Status verified 2018-03

CONDITIONS: Unrecognized Condition
Keywords: Transplant renal artery stenosis; Endovascular repair; Post-operative outcome
MeSH Terms: interventions — Angioplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Angioplasty for Transplant Renal Artery Stenosis (TRAS) — The angioplasty is an endovascular treatment for artery stenosis, which could be associated with stenting or not.
  Other Names: Endovascular treatment

SUMMARY:
Stenosis of the renal graft arteries occurs in 1 to 26% of cases and can damage the graft. Endovascular treatment is first-line treatment. The main objective of this study is to identify the predictive factors of failure of peri-anastomotic.

DETAILED DESCRIPTION:
The aim of this study was to evaluate the post-operative outcomes following endovascular treatment of TRAS (Transplant Renal Artery Stenosis).

This retrospective, monocentric study included patients with peri-anastomotic stenosis of the renal graft from 2000 to 2017. The stenosis is defined by a reduction of at least 50% of the arterial diameter during arteriography. Technical success was defined as residual stenosis less than 30% of the arterial diameter after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* All patients who had a renal transplant from brain-dead donors or from living donors
* All patients who had a Transplant Renal Artery Stenosis

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This retrospective, monocentric study included patients with peri-anastomotic stenosis of the renal graft from 2000 to 2017.
Sampling Method: Non-Probability Sample
Enrollment: 1323 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
The technical success rate of endovascular treatment | 30 days
  The stenosis is defined by a reduction of at least 50% of the arterial diameter during arteriography. Technical success was defined as residual stenosis less than 30% of the arterial diameter after the procedure

SECONDARY OUTCOMES:
Morbidity rate | 30 days
  Morbidity rate is defined as the development of post-operative complications. Minor and major complications are recorded, corresponding to Clavien Dindo classification
Mortality rate | 30 days
  All death are recorded to identify the mortality rate

IPD SHARING:
Plan to Share IPD: No
Submission at several congress: WCE2017, AFU2017 Publication at the Journal of Urology in March 2018